CLINICAL TRIAL: NCT03938415
Title: Acupuncture for Vasectomy Pre-procedural Anxiety and Pain Control in the Primary Care Setting: A Randomized Comparative Effectiveness Trial
Brief Title: Acupuncture for Vasectomy Pre-procedural Anxiety and Pain Control in the Primary Care Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Matthew Snyder (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Matthew Snyder, Principal Investigator, Mike O'Callaghan Military Hospital
Organization: Mike O'Callaghan Military Hospital (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FWH20190062H
Record Dates: First submitted 2019-04-30; First posted 2019-05-06 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Acupuncture; Pain, Postoperative; Vasectomy
MeSH Terms: conditions — Pain, Postoperative | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture (Experimental): Acupuncture
  Interventions: Procedure: Acupuncture
- Standardized pre-procedure medications (Active Comparator): The clinic standardized pre-procedure medications alone
  Interventions: Other: Standardized pre-procedure medications

INTERVENTIONS:
Procedure: Acupuncture — Acupuncture involving the Koffman protocol (body acupuncture) for anxiety control (needles will be placed at bilateral LR-3, bilateral LI-4, GV 24.5 and GV 20) and Auricular ATP Plus (ear) for pain control (needles will be placed at points hippocampus, amygdala, hypothalamus, prefrontal cortex, Point Zero, Shen Men, vagus, insula, external genitalia). Subjects who tolerate the auricular needles will be offered replacement with ASP acupuncture needles for continued pain management post-procedure. The subjects will receive local anesthetic during the vasectomy per standardized clinic protocol.
  Arms: Acupuncture
Other: Standardized pre-procedure medications — The clinic standardized pre-procedure medications alone (which include diazepam 5 mg by mouth (PO) x1 30 minutes prior to the procedure, an additional 5 mg PO x1 15 minutes later if desired effect is not achieved; and oxycodone/acetaminophen 5/325 mg PO x 1 30 minutes prior to the procedure. The subjects will receive local anesthetic during the vasectomy per standardized clinic protocol.
  Arms: Standardized pre-procedure medications

SUMMARY:
This study compares auricular (ear) acupuncture and body acupuncture (Koffman protocol) versus clinic standardized pre-vasectomy medications to determine which has better outcomes at improving pre-procedural anxiety and procedural pain relief and medication usage in adult male patients following vasectomy.

DETAILED DESCRIPTION:
The investigators will compare auricular (ear) and body acupuncture (Koffman protocol) versus clinic standardized pre-vasectomy medications to determine which has better outcomes at improving pre-procedural anxiety and procedural pain relief and medication usage in adult male patients following vasectomy. In this efficacy trial, the investigators hypothesize that acupuncture will provide therapeutic anxiety and pain relief during and after vasectomy. The investigators will measure anxiety immediately before and prior to the procedure and before and after the intervention via a standardized anxiety scale (comparative). The investigators will also measure pain control immediately after the procedure using Defense and Veterans Pain Rating Scale (DVPRS). At the post op check (2-4 days after procedure) subjects will fill out a patient satisfaction survey. During the recovery period over 2 weeks, a medication usage diary will be kept by the subject including the time when the patient returns to full duties.

ELIGIBILITY:
**Patients must be able to get care at Nellis Air Force Base (a military installation) in order to participate in this study**

Inclusion Criteria:

* Male active duty members and DoD beneficiaries aged 25 years or older
* Scheduled for a vasectomy

Exclusion Criteria:

* Repeat vasectomy
* Chronic pain medication/benzodiazepine use
* Current pain contract/pain management
* Current anxiolytic medication
* History of needle shock
* Diagnosis of anxiety
* Needle phobia
* Blood/injury phobia
* History of vasovagal reflex response

Min Age: 25 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2025-04-11 (Actual); Study Completion 2025-04-11 (Actual)

PRIMARY OUTCOMES:
Change in Hospital Anxiety and Depression Scale (HADS) -- Medication Arm | Day 0 (2x)
  The HADS is a self-rating scale developed to assess psychological distress in non-psychiatric patients. It consists of two subscales, Anxiety and Depression, each having seven items and a score range of 0 to 21. The HADS has been satisfactorily used in the general population and a number of clinical settings. A score less than 8 is considered as being normal, 8 to 10 as suggestive of anxiety or depression, and greater than 11 as being probable of anxiety or depression. The HADS score is ordinal and will be analyzed using nonparametric methods
Change in Hospital Anxiety and Depression Scale (HADS) -- Acupuncture Arm | Day 0 (2x)
  The HADS is a self-rating scale developed to assess psychological distress in non-psychiatric patients. It consists of two subscales, Anxiety and Depression, each having seven items and a score range of 0 to 21. The HADS has been satisfactorily used in the general population and a number of clinical settings. A score less than 8 is considered as being normal, 8 to 10 as suggestive of anxiety or depression, and greater than 11 as being probable of anxiety or depression. The HADS score is ordinal and will be analyzed using nonparametric methods
Change in Defense and Veterans Pain Rating Scale (DVPRS) | Day: 0 (pre-procedure), 0 (post-procedure),1,2,3,4,5,6,7,8,9,10,11,12,13,14
  The DVPRS consists of an 11-point numerical rating scale with 0 indicating no pain and 10 indicating severe pain. It has been confirmed for reliability and validity in measuring both acute and chronic pain, and is currently the standard for pain measurement throughout DoD and VA health systems. The DVPRS has demonstrated linear scale qualities allowing parametric methods to be used

CONTACTS AND LOCATIONS:
Locations (1):
- Mike O'Callaghan Military Medical Center, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No
The investigators do not plan on sharing data

REFERENCES:
- [Background] Wunsch JK, Klausenitz C, Janner H, Hesse T, Mustea A, Hahnenkamp K, Petersmann A, Usichenko TI. Auricular acupuncture for treatment of preoperative anxiety in patients scheduled for ambulatory gynaecological surgery: a prospective controlled investigation with a non-randomised arm. Acupunct Med. 2018 Aug;36(4):222-227. doi: 10.1136/acupmed-2017-011456. Epub 2018 Jul 9. PMID 29986900
- [Background] Wang SM, Peloquin C, Kain ZN. The use of auricular acupuncture to reduce preoperative anxiety. Anesth Analg. 2001 Nov;93(5):1178-80, table of contents. doi: 10.1097/00000539-200111000-00024. PMID 11682391
- [Background] Wang SM, Maranets I, Weinberg ME, Caldwell-Andrews AA, Kain ZN. Parental auricular acupuncture as an adjunct for parental presence during induction of anesthesia. Anesthesiology. 2004 Jun;100(6):1399-404. doi: 10.1097/00000542-200406000-00011. PMID 15166558
- [Background] Thomas M, Eriksson SV, Lundeberg T. A comparative study of diazepam and acupuncture in patients with osteoarthritis pain: a placebo controlled study. Am J Chin Med. 1991;19(2):95-100. doi: 10.1142/S0192415X91000156. PMID 1816730
- [Background] Sinha V, Ramasamy R. Post-vasectomy pain syndrome: diagnosis, management and treatment options. Transl Androl Urol. 2017 May;6(Suppl 1):S44-S47. doi: 10.21037/tau.2017.05.33. PMID 28725617

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-04-04): https://cdn.clinicaltrials.gov/large-docs/15/NCT03938415/Prot_SAP_000.pdf
  • Informed Consent Form (2019-01-22): https://cdn.clinicaltrials.gov/large-docs/15/NCT03938415/ICF_001.pdf